CLINICAL TRIAL: NCT01686789
Title: Randomized Controlled Open Label Trial of Peg Alpha 2a Interferon and Adjusted-dose of Ribavirin vs. Standard Therapy in the Treatment of Naive Chronic Hepatitis C Patients Infected With Genotype 4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Abdulaziz Medical City (Other Government)
Responsible Party: Principal Investigator, Faisal M Sanai, Consultant Hepatologist & Liver Transplant Physician, King Abdulaziz Medical City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC08-064
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pegylated interferon alpha-2a plus standard dose ribavirin (Active Comparator): Pegylated interferon alpha-2a 180 mcg weekly plus standard dose ribavirin 100-1200 mg/day for 48 weeks
  Interventions: Drug: Pegylated interferon alpha-2a
- Pegylated interferon alpha-2a 180 mcgs adjusted dose ribavirin (Experimental): Pegylated interferon alpha-2a 180 mcg weekly plus adjusted dose ribavirin for 48 weeks
  Interventions: Drug: Pegylated interferon alpha-2a

INTERVENTIONS:
Drug: Pegylated interferon alpha-2a

SUMMARY:
The study aims to study the outcome of pharmacokinetics-adjusted dose ribavirin (plus pegIFN) on the SVR in chronic HCV patients.

DETAILED DESCRIPTION:
Background: The introduction of Peg interferon and Ribavirin (an oral nucleoside analogue) for chronic Hepatitis C has led to the concept that chronic hepatitis C (HCV) is a curable disease. Improvement of treatment efficacy is still a major challenge. Optimal Ribavirin doses are essential to achieve SVR (sustained virological response). A recent trial showed significantly higher sustained virological response (SVR) in patients receiving 15.2 mg/kg/day of Ribavirin compared with 13.3 mg/kg/day. Ribavirin was given in combination with Peg interferon alpha-2b (1). A small pilot study, in which 10 patients with Chronic Hepatitis C genotype 1 were treated with Ribavirin dosage up to 3600 mg/day- mean of 2540 mg/day- plus Peg-interferon alpha-2a, achieving a target concentration of Ribavirin >15 micromol before W 12, led to 90% of SVR(2). All patients managed to complete the one year treatment period but all needed EPO and two were transfused.

Patient's global exposure to Ribavirin as evaluated by the area under the curve (AUC) seems more pertinent in terms of exposure-effect relationship than measuring Ribavirin level at any single time point. A recent study showed in HCV patients infected with genotype 1 that Ribavirin plasma exposure after the first dose (i.e., interdose AUC0-12h or abbreviated AUC0-4h) was significantly and strongly linked with SVR, whereas AUCs determined at W12 and W24 and trough concentrations at Day 0 and W12 were not (3).

Therefore, we propose a randomized controlled trial to investigate whether adjusted Ribavirin doses based on AUC0-4h obtained at D-7 after 600mg dose of Ribavirin versus fixed standard doses can improve outcome in treatment of chronic hepatitis C naïve patients infected with genotype 4.

Methodology: After AUC0-4h has been determined at D-7 (7 days before randomization) for 190 genotype 4 patients recruited into the trial, the patients are randomized into two groups: Group A: to receive standard dose of Ribavirin 1000-1200 mg/day) and Group B: to receive adjusted-dose of Ribavirin according to AUC0-4h. The individual calculated dose should be administered for each patient beginning on the first day of treatment. Both groups will receive combination treatment with peginterferon alpha 2a 180 mcg/week for a total of 48 weeks.

Both treatment groups will receive Darbepoetin if subsequent Hb is < 11 g/dl for males and females. Our main inclusion criteria will be: patients 18-70 years old with serological evidence of chronic hepatitis C and positive HCV RNA of genotype 4, with a liver biopsy within 3 years prior to recruitment. Our main exclusion criteria will be: decompensated cirrhotic patients, HBV/HIV co-infection, evidence of hepatocellular carcinoma (HCC), significant evolutive cardiovascular, pulmonary, renal or psychiatric disease, pregnancy/breast feeding or patients post liver transplantation and anemia.

Our primary outcome will be: HCV-RNA negativity 24 weeks after the end of treatment (SVR) (input adjusted dose on SVR). Our secondary outcome will be: rapid virological response (RVR), early virological response (EVR), partial early virological response (pEVR), end of treatment response (ETR), relapse after (ETR), biochemical response and safety and tolerability of high doses of Ribavirin.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years of age
2. Chronic hepatitis C documented by a detectable HCV RNA level by a PCR performed within 3 months -A liver biopsy performed within 3 years or fibro test/fibroscan within 1 year of inclusion.
3. Naive patients
4. Genotype 4
5. Compensated cirrhosis hepatitis C liver disease (Child-Pugh ≤ 6)
6. Patient needing, according to the physician, the initiation of a combined therapy of pegylated interferon alfa plus Ribavirin
7. Negative HBsAg test and HIV-Elisa test
8. Negative pregnancy test at baseline in women in age of procreation
9. Efficient contraception all along the treatment period, and for 6 months after discontinuation of the treatment for women and men

Exclusion Criteria:

1. Decompensated Cirrhotic patients
2. HBV or HIV co-infection
3. Evidence of hepatocellular carcinoma
4. Significant and evolutive cardiovascular, pulmonary, severe psychiatric disorder or renal dysfunction (calculated creatinine CL < 50 ml/min) *. Patients who met the trial criteria if subsequent calculated creatinine CL < 50 ml/min may need ribavirin dose reduction.
5. Non compensated thyroid dysfunction
6. Recent history of epilepsy (less than 6 months)
7. Absolute contraindications to one of the drug of combination therapy
8. Any non-compensated cardiac disease including ischemic heart disease Chronic cardiac failure (grade III or IV - NYHA classification)
9. Uncontrolled high blood pressure (SBP > 180 mmHg during inclusion in spite of hypertension treatment)
10. Pregnancy or breast feeding.
11. Post liver transplantation patient with HCV
12. Alcohol or drug induced liver disease.
13. Metabolic or autoimmune liver disease.
14. Hemoglobinopathies or anemia; hemoglobin <12 gm /dl for females and <12.5 for males not corrected by erythropoietin
15. Neutropenia (<1500/mm³)
16. Thrombocytopenia (<90,000/mm3), thrombocytosis (> 500,000/mm3)
17. Patients with evolutive diabetic or hypertensive retinopathy. Patients who are stable can be included but should be regularly followed during treatment.
18. Hypersensitivity to epoetin beta or one of its excipients
19. Previous history or increased risk of venous thrombosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2011-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Sustained virological response | 72 weeks
  Detectability of HCV RNA after 24 weeks of treatment completion by a realTime PCR-based technique

SECONDARY OUTCOMES:
Requirement of blood-related products | 48 weeks
  The development of anemia or requirement of blood-related products

CONTACTS AND LOCATIONS:
Locations (3):
- Saudi Arabia (3):
  - King Faisal Specialist Hospital & Research Centre, Riyadh
  - King Abdulaziz Medical City, Riyadh
  - King Khaled University Hospital, Riyadh